CLINICAL TRIAL: NCT01000363
Title: Diabetes Medical Group Visits Pilot Study
Brief Title: Diabetes Group Visits
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Johnson & Johnson (Industry); American Association of Diabetes Educators (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Other Study IDs: IRB00029165
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spanish speaking group: Diabetes medical group visits will be held at the Grady North DeKalb satellite clinic the third Thursday of the month starting in October 2009. There will be two cohorts of patients- English speaking patients and Spanish speaking patients. Each group will be scheduled for 4 2-hour group visits throughout a period of 9 months. These visits will be every 8 weeks for each group. During the visit, the patient will be seen by a physician, attend a diabetes education session, re-fill their diabetes medications, get orders for labs due, vaccinations and diabetes-related referrals.
- English speaking group: Each group will be scheduled for 4 2-hour group visits throughout a period of 9 months. These visits will be every 8 weeks for each group. During the visit, the patient will be seen by a physician, attend a diabetes education session, re-fill their diabetes medications, get orders for labs due, vaccinations and diabetes-related referrals.
  This visit will only focus on the patient's diabetes care. Each patient will continue to see their regular physician for their health care.
  All of the services that will be provided at the medical group visit are standard of care and are the same that the patient will receive in a one-on-one visit. However, this format will allow the patient to been seen by the physician and receive diabetes education in one visit.

SUMMARY:
This pilot study aims to increase access to diabetes education by delivering it in a culturally-appropriate community setting and by involving different members of the diabetes care team including physicians, diabetes educators, and health promoters/community health workers.

Diabetes medical group visits will be held at the Grady North DeKalb satellite clinic the third Thursday of the month starting in October 2009. There will be two cohorts of patients- English speaking patients and Spanish speaking patients. Each group will be scheduled for 4 2-hour group visits throughout a period of 9 months. These visits will be every 8 weeks for each group. During the visit, the patient will be seen by a physician, attend a diabetes education session, re-fill their diabetes medications and receive lab orders.

DETAILED DESCRIPTION:
Patients who participate in the diabetes group visits should achieve improvement in Clinical outcomes - better A1C levels, reduced blood pressure, reduced cholesterol levels ; adherence to evidence-based medicine - keeping appointments and scheduling eye exams, foot-checks, and/or taking medication as prescribed; behavioral outcomes- goal setting, achievement of goals, problem solving; access - attendance at educational sessions; ability to obtain affordable medications and devices; and satisfaction among patients and health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Primary care at the Grady North DeKalb Health center
* Valid Grady card
* Age 18-80
* HbA1c>=8.0% - 11.0%
* Must speak English or Spanish

Exclusion Criteria:

* -Primary care provider excludes patient from study
* Patient is reluctant to participate in a group visit
* Reduced life expectancy as determined by any of the following:
* End-stage renal disease on dialysis
* Active congestive heart failure II and IV
* Lung disease requiring supplemental oxygen
* Current malignancy with any evidence of disease or currently undergoing chemotherapy or radiation therapy
* Cirrhosis of the liver
* AIDS
* Mayor mental health disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to study a total of 40 patients with a known history of type 1 or type 2 diabetes, ages 18-80. Patients included within this study will be determined by the set of inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patients who participate in the diabetes group visits should achieve improvement in Clinical outcomes - better A1C levels, reduced blood pressure, reduced cholesterol levels | 1 year

SECONDARY OUTCOMES:
keeping appointments and scheduling eye exams, foot checks | 1 year
goal setting, achievement of goals, problem solving; access | 1 year
attendance at educational sessions; and satisfaction among patients and health professionals | 1 year
behavioral outcomes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — EUSOM
Locations (1):
- Grady North DeKalb Clinic, Chamblee, Georgia, United States